CLINICAL TRIAL: NCT05917457
Title: Investigation of the Effects of Balance Coordination and Reinforcement Training on Gait, Mobility and Posture in Children with Low Vision
Brief Title: Investigation of the Effects of Balance Coordination and Strengthening Training on Gait, Mobility and Posture in Children with Low Vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Server ERDOĞMUŞ, Physiotherapist Server ERDOĞMUŞ, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Children with Low Vision
Record Dates: First submitted 2023-05-29; First posted 2023-06-23 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Children with Low Vision
Keywords: Low vision; visually impaired; balance; strength training; walking
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Intervention Model Description: Criteria for Inclusion of Volunteers in the Study and Control Group in the Research:
  to be in the age of 7-14, Except for visual impairment (neurological and systemic diseases, hearing impairment, etc. ) not having an additional disease October, Having been diagnosed with low vision, To be able to establish cooperation, Volunteering to participate in the study The 25 individuals who met the inclusion criteria were divided into 2 groups, including 13 in the study group and 12 in the control group
Masking Description: they knew which groups they were in and the researcher knew where they were too.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental): to be in the age of 7-14, Except for visual impairment (neurological and systemic diseases, hearing impairment, etc. ) not having an additional disease Having been diagnosed with low vision, To be able to establish cooperation, Volunteering to participate in the study 12 children with these criteria
  Interventions: Other: balance coordination and strengthening training
- control group (No Intervention): to be in the age of 7-14, Except for visual impairment (neurological and systemic diseases, hearing impairment, etc. ) not having an additional disease, Having been diagnosed with low vision, To be able to establish cooperation, Volunteering to participate in the study 10 children with these criteria

INTERVENTIONS:
Other: balance coordination and strengthening training — The 25 individuals who met the inclusion criteria were divided into 2 groups, including 13 in the study group and 12 in the control group.
  Study group: Low vision children were given balance, coordination training and general strengthening training with sandbags for 70 minutes 3 days a week (5-minute warm-up phase, 20-minute balance training, 20-minute coordination training, 20-minute strengthening training and 5-minute cooling phase) for 8 weeks.
  Arms: treatment group

SUMMARY:
The aim of this research is to examine and evaluate the effects of balance coordination and strengthening training on gait, mobility and posture in children with low vision

The hypotheses of our study:

H1: Balance coordination and strengthening training has an effect on gait, mobility and posture in children with low vision.

H2: Balance coordination and strengthening training has no effect on gait, mobility and posture in children with low vision.

DETAILED DESCRIPTION:
The aim of this study is to examine and evaluate the effects of balance coordination and strengthening training on gait, mobility and posture in children with low vision.

A total of 22 low-vision individuals were included in the study. Individuals were randomly divided into two groups as Control (n=10) and Study (n=12). The treatment group received 70 min balance (20 min), coordination (20 min) and strengthening (20 min) training 3 days a week for 8 weeks. No additional treatment was applied to the control group. Evaluations were performed before treatment and at the end of 8 weeks.

In the evaluations; Bruininks-Oseretsky Motor Proficiency Test 2 Short Form (BOT2- KF), New York Posture Analysis, Manual November muscle strength assessment, G-Walk Gait Analysis, Independent Mobility Questionnaire (BMA) were used.

ELIGIBILITY:
Inclusion Criteria:

* To be in the age December of 7-14,
* Except for visual impairment (neurological and systemic diseases, hearing impairment, etc. ) not having an additional disease,
* Having been diagnosed with low vision,
* To be able to establish cooperation,
* Volunteering to participate in the study

Exclusion Criteria:

* Not being diagnosed with low vision,
* Except for visual impairment (neurological and systemic diseases, hearing impairment, etc. ) having an additional disease,
* Not volunteering to participate in the study

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of motor competence | 8 weeks
  The Bruininks- Oseretsky Motor Proficiency Test Short Form was used to evaluate motor competence in the cases.
posture analysis | 8 weeks
  New York Posture Analysis was used to evaluate postures of the cases.
muscle strength assessment | 8 weeks
  The Lovett method was used for the muscle strength
Evaluation of Walking Parameters | 8 weeks
  G-Walk system was used
Mobility Level Assessment | 8 weeks
  Independent Mobility Questionnaire (IMQ) was used

CONTACTS AND LOCATIONS:
Overall Officials: ERDOĞAN KAVLAK, Study Director — Pamukkale University
Locations (1):
- Kınıklı Campus, Üniversite St. No:11 20160 Pamukkale / DENİZLİ, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
1. Treatment group: Children with low vision will be given balance, coordination training and strengthening with sandbags for 75 minutes 3 days a week, for 8 weeks.
  2. Control Group: No training will be given except for evaluations.
Supporting Information: Study Protocol, ICF
Time Frame: July 2022-June 2023